CLINICAL TRIAL: NCT04669405
Title: The Effectiveness of High Intensity Laser Therapy in the Treatment of Hemiplegic Shoulder Pain: A Prospective Randomized Controlled Study
Brief Title: High Intensity Laser Therapy in the Treatment of Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7
Record Dates: First submitted 2020-12-14; First posted 2020-12-16 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hemiplegia
Keywords: hemiplehic shoulder pain; rotator cuff tear; high intensity laser therapy; exercise; ultrasound
MeSH Terms: conditions — Hemiplegia; Rotator Cuff Injuries; Motor Activity | interventions — Rehabilitation; Exercise Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT group (Active Comparator): Patients with hemiplegic shoulder pain with partial thickness rotator cuff receiving high intensity laser therapy.
  Interventions: Device: High intensity laser therapy; Other: Therapeutic Exercise
- Control group (Other): Patients with hemiplegic shoulder pain with partial thickness rotator cuff receiving exercise.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Device: High intensity laser therapy — A prospective, randomized, controlled study was undertaken. A total of 44 patients who met inclusion criteria were randomly divided into two groups. HILT group (n=22) received 3 sessions of HILT per week for 3 weeks in addition to the multidisciplinary stroke rehabilitation and exercise program which performed 5 sessions per week for 3 weeks. Control group (n=22) received a multidisciplinary stroke rehabilitation and exercise program for HSP of 5 sessions per week for 3 weeks.
  Other Names: Rehabilitation program
  Arms: HILT group
Other: Therapeutic Exercise — A prospective, randomized, controlled study was undertaken. A total of 44 patients who met inclusion criteria were randomly divided into two groups. HILT group (n=22) received 3 sessions of HILT per week for 3 weeks in addition to the multidisciplinary stroke rehabilitation and exercise program which performed 5 sessions per week for 3 weeks. Control group (n=22) received a multidisciplinary stroke rehabilitation and exercise program for HSP of 5 sessions per week for 3 weeks.
  Other Names: Rehabilitation program

SUMMARY:
High intensity laser therapy (HILT) has been considered as a treatment option for shoulder pain. To our knowledge, the effectiveness of HILT in patients with hemiplegic shoulder pain (HSP) with partial thickness rotator cuff tear (PTRCT) is unknown. In this study, we intended to investigate the effectiveness of HILT on pain, disability, function and quality of life in patients with HSP accompanied by PTRCT.

DETAILED DESCRIPTION:
The study was designed as prospective, randomized, controlled trial. Patients with HSP accompanied by PTRCT (n=44) were randomly assigned to HILT and control groups. Group 1 (HILT group, n=22) received 3 sessions of HILT per week for 3 weeks in addition to the exercise program which performed 5 sessions per week for 3 weeks. Group 2 (Control group, n=22) received an exercise program for HSP of 5 sessions per week for 3 weeks.

Participants were evaluated with Visual Analog Scale (VAS), passive Range of Motion (ROM), Shoulder Pain and Disability Index (SPADI), Nottingham Health Profile (NHP), Functional Independence Measure (FIM) and ultrasonographic PTRCT size.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HSP (at least 4/10 points from VAS) aged 18-75 years with hemiplegia duration> 6 months, suffered a stroke resulting in unilateral hemiplegia for the first time, and who had partial thickness RCT after ultrasonographic evaluation due to shoulder pain

Exclusion Criteria:

* Cases who had inflammatory rheumatic disease, cervical radiculopathy, diabetes mellitus, thyroid disease, coronary heart disease, cardiac pace-maker, neurological disease, shoulder surgery, and shoulder injection in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Pain of the hemiplegic shoulder | Through study completion, an average of 3 weeks (Change from baseline hemiplegic shoulder pain of the patients at 3 weeks
  Severity of pain was assessed using the standart 10 cm VAS with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end

SECONDARY OUTCOMES:
Range of motion (ROM) of the hemiplegic shoulder | Through study completion, an average of 3 weeks (Change from baseline hemiplegic shoulder ROM of the patients at 3 weeks
  Passive ROM measurements of shoulder external rotation, abduction, and flexion movements were recorded by a universal goniometer.
Shoulder functional status (SPADI) | Through study completion, an average of 3 weeks (Change from baseline hemiplegic shoulder functional status of the patients at 3 weeks
  SPADI is self-administered questionnaire composed of 5 items assessing pain and 8 items assessing disability. The score varied from 0% to 100%, with higher scores reflected greater pain and disability
Motor recovery | Through study completion, an average of 3 weeks (Change from baseline hemiplegic arm motor recovery of the patients at 3 weeks
  Brunnstrom Recovery Stage (BRS) was used to appreciated the motor function level in the patients. The recovery are divided into six stages: In the 1st stage, there is complete flaccidity, and no voluntary movements in the involved body area, while the 6th stage indicates normal function
Spastisity | Through study completion, an average of 3 weeks (Change from baseline hemiplegic arm spasticity of the patients at 3 weeks
  The five-point Modified Ashworth Scale (MAS), a clinical scale ranging from 0 to 4 (0 being normal muscle tone, and 4 being rigid) was used for measuring spasticity and muscle tone.
Functional status (FIM) | Through study completion, an average of 3 weeks (Change from baseline functional status of the patients at 3 weeks
  FIM is a universal assessment tool consisting of a total of 18 items that explores an individual's several physical and social functions, such as self-care, transfer, locomotion, sphincter control, communication and social cognition. Each item is scored on a 7-point ordinal scale ranging from complete independence (score= 7) to complete dependence (score= 1). Higher FIM scores indicate higher levels of independence
Quality of life of the hemiplegic patient | Through study completion, an average of 3 weeks (Change from baseline quality of life of the patients at 3 weeks
  Nottingham Health Profile (NHP), a life quality test, includes 38 yes / no statements regarding pain, physical mobility, emotional reactions, sleep, social isolation and energy level. Ratings on each component are weighted to give a score between 0 and 100. Higher NHP scores show a higher level of trouble
Rotator cuff tear size | Through study completion, an average of 3 weeks (Change from baseline rotator tear cuff size of the patients at 3 weeks
  Ultrasonographycally detected a hypoechoic / anechoic focus in the cuff material or a hypoechoic / anechoic defect in the tendon that holds the bursal or articular surface

CONTACTS AND LOCATIONS:
Overall Officials: Evren Yaşar, MD, Study Director — Health Sciences University, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital; Nurdan Korkmaz, MD, Principal Investigator — Health Sciences University, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Korkmaz N, Gurcay E, Demir Y, Tezen O, Korkmaz I, Atar MO, Yasar E. The effectiveness of high-intensity laser therapy in the treatment of post-stroke patients with hemiplegic shoulder pain: a prospective randomized controlled study. Lasers Med Sci. 2022 Feb;37(1):645-653. doi: 10.1007/s10103-021-03316-y. Epub 2021 Apr 8. PMID 33829317